CLINICAL TRIAL: NCT01283152
Title: Randomized Controlled Trial Evaluating the Efficacy of Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) in Patients With Hepatic Encephalopathy.
Brief Title: Efficacy Study of Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) Versus Lactulose in Patients With Hepatic Encephalopathy.
Acronym: PSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Rahimi, MD, MSCR, MD, MSCR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 072010-121
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Hepatic Encephalopathy; Cirrhosis; Portosystemic Encephalopathy; PSE
Keywords: Hepatic Encephalopathy; HE; Cirrhosis; PSE; Portosystemic Encephalopathy; Hepatic coma; AMS; Altered mental status; Complications of cirrhosis; Chronic liver disease
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Golytely; polyethylene glycol 3350; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyethylene glycol 3350-electrolyte solution (GoLYTELY®) (Active Comparator)
  Interventions: Drug: Polyethylene glycol 3350-electrolyte solution (GoLYTELY®)
- Lactulose (Other): Per standard of care
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Polyethylene glycol 3350-electrolyte solution (GoLYTELY®) — If randomized to this arm, subjects will receive a 1 time dose of 1 gallon
  Other Names: GoLYTELY® or Miralax®
  Arms: Polyethylene glycol 3350-electrolyte solution (GoLYTELY®)
Drug: Lactulose — If randomized to this arm, subjects will receive 10-30 grams per standard of care
  Arms: Lactulose

SUMMARY:
This study is being done to find out if the laxative polyethylene glycol (also known as GoLYTELY® or Miralax®) can treat your hepatic encephalopathy (confusion due to your liver disease and/or cirrhosis) better and/or more safely than lactulose (another laxative). In this study, the investigators will evaluate if polyethylene glycol (GoLYTELY®) is more effective than lactulose on neurocognition (memory and thinking skills) and determine if it decreases the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-80
2. Male and female subjects of all races and ethnicities including Spanish speaking subjects
3. Cirrhosis of any cause
4. Any grade of hepatic encephalopathy (1-4)
5. A legally authorized representative has to be able and willing to comply with all protocol procedures and to understand, sign and date an informed consent document, and authorize access to protected health information on the subjects behalf

Exclusion Criteria:

1. Acute liver failure
2. Structural brain lesions (as indicated by computed tomography imaging if available and confirmed by neurological exam)
3. Other causes of altered mental status (i.e. not meeting the definition of hepatic encephalopathy)
4. Previous use of rifaximin or neomycin in past 7 days
5. Prisoners
6. Pregnancy
7. <18 years old
8. Serum sodium <125 mEq/L
9. Receiving > 1 dose of lactulose prior to enrollment
10. Uncontrolled infection with hemodynamic instability requiring vasopressors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Rahimi, MD, MSCR, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center and Parkland Memorial Health and Hospital System, Dallas, Texas, United States

REFERENCES:
- [Background] Doran AE, Shah NL. Polyethylene glycol for hepatic encephalopathy: a new solution to purge an old problem? JAMA Intern Med. 2014 Nov;174(11):1734-5. doi: 10.1001/jamainternmed.2014.3501. No abstract available. PMID 25244573
- [Result] Rahimi RS, Singal AG, Cuthbert JA, Rockey DC. Lactulose vs polyethylene glycol 3350--electrolyte solution for treatment of overt hepatic encephalopathy: the HELP randomized clinical trial. JAMA Intern Med. 2014 Nov;174(11):1727-33. doi: 10.1001/jamainternmed.2014.4746. PMID 25243839
- See also: PubMed link to abstract — http://www.ncbi.nlm.nih.gov/pubmed/25243839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized clinical trial was performed at Parkland Memorial Hospital, Dallas, Texas, from January 2011 to June 2012. All patients presenting to the emergency department with known cirrhosis and altered mental status (AMS) were eligible.
Pre-assignment Details: A total of 186 patients were screened; 50 eligible patients were randomized to standard-of-care treatment (lactulose) or PEG. The most common reasons for exclusion were that the patient had received more than 1 dose of lactulose in the emergency department prior to consent, that a LAR was not available, or that the patient did not have HE.
Period: Overall Study
Arm/Group | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) | Lactulose
Started | 25 | 25
ITT Population | 25 | 25
Study Treatment Received | 25 | 25
24-hr HESA Attempted | 25 | 25
Completed | 23 | 25
Not Completed | 2 | 0
Not completed — Discharged prior to 24 hr assessment | 1 | 0
Not completed — Refused HESA | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) | Lactulose | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7) | 56 (11) | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 2 | 2 | 4
  Asian | 1 | 0 | 1
  White, Hispanic | 20 | 15 | 35
  White, non-Hispanic | 2 | 8 | 10
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Cirrhosis cause [Number; unit: participants]
  Alcoholic Liver Disease | 10 | 9 | 19
  Cryptogenic | 6 | 6 | 12
  Hepatitis C | 8 | 9 | 17
  Hepatitis B | 1 | 1 | 2
White Blood Cell count [Mean (Standard Deviation); unit: cells*10^9/L] | 6.3 (2.6) | 6.2 (2.6) | 6.2 (2.6)
Blood Lab Values [Mean (Standard Deviation); unit: mg/dL]
  Blood Urea Nitrogen | 30 (17) | 21 (11) | 26 (15)
  Creatinine | 1.7 (1.29) | 1.12 (0.52) | 1.41 (1.02)
  Total Bilirubin | 3.6 (3) | 2.9 (1.4) | 3.3 (2.3)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: unitless (ratio)] — INR is based on the ratio of the patient's prothrombin time and the normal mean prothrombin time.
  unitless (ratio) | 1.5 (0.4) | 1.4 (0.3) | 1.5 (0.4)
Albumin [Mean (Standard Deviation); unit: g/dL] | 2.7 (0.6) | 2.8 (0.5) | 2.7 (0.6)
MELD and CTP Scores [Mean (Standard Deviation); unit: units on a scale] — Model of End-stage Liver Disease (MELD) score assesses the severity of chronic liver disease. MELD has a range from less than 9 to more than 40 with higher numbers indicating greater severity; Child-Turcotte-Pugh (CTP) score assesses the prognosis of chronic liver disease. CTP has a range from 5 to 15 with higher numbers indicating a worse prognosis.
  units on a scale
    MELD score | 17 (6) | 17 (5) | 17 (5)
    CTP score | 10 (2) | 10 (1) | 10 (2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Improvement of 1 or More in HE Grade at 24 Hours
Description: Hepatic Encephalopathy Scoring Algorithm (HESA) at the 24 hour time point of when the subject was recruited (HESA improvement by at least 1 grade). HESA ranges from 0 to 3, with higher numbers indicating a more severe grade of hepatic encephalopathy. Study will continue at every 24 hour time point until the subject achieves his or her baseline mental state and/or grade 0 based on the HESA
Time Frame: Baseline to 24 hours
Population: All participants who completed the study
Measure: Number; unit: participants
Arm/Group | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) | Lactulose
Number analyzed (Participants) | 23 | 25
participants | 21 | 13

2. Secondary Outcome: Hospital Duration/Length of Stay
Time Frame: From time of admission to time of discharge or death
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) | Lactulose
Number analyzed (Participants) | 25 | 25
days | 4 (3) | 8 (12)

3. Primary Outcome: Change in HE Grade at 24 Hours
Description: Hepatic Encephalopathy Scoring Algorithm (HESA) at the 24 hour time point of when the subject was recruited. HESA ranges from 0 to 3, with higher numbers indicating a more severe grade of hepatic encephalopathy. Study will continue at every 24 hour time point until the subject achieves his or her baseline mental state and/or grade 0 based on the HESA
Time Frame: Baseline to 24 hours
Population: All participants who completed the study
Measure: Number; unit: participants
Arm/Group | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) | Lactulose
Number analyzed (Participants) | 23 | 25
participants
  improvement of 1 HESA grade | 10 | 9
  improvement of 2 HESA grades | 9 | 3
  improvement of 3 HESA grades | 1 | 1
  No HESA improvement | 2 | 12
  HESA grade 0 at 24 hours | 10 | 2

ADVERSE EVENTS:
Arm/Group | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) | Lactulose
Serious Adverse Events (participants affected / at risk) | 3/25 | 5/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyethylene Glycol 3350-electrolyte Solution (GoLYTELY®) (N=25) | Lactulose (N=25)
Death (Cardiac disorders) | 0 (0) | 2 — Cardiorespiratory---not related
Death (Gastrointestinal disorders) | 1 | 0 (0) — Hemoperitoneum--Not related
Recurrent HE (Gastrointestinal disorders) | 2 | 1 — Possibly study related
Intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 — Probably not related
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 — Probably not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No